CLINICAL TRIAL: NCT01805674
Title: Study to Evaluate the Changes in Quality of Life in Menopausal Women After the Administration of Soy Isoflavones Combined With Magnolia Extract
Brief Title: Isoflavones and Magnolia Extract in the Quality of Life in Menopausal Women
Acronym: ESTROCALVI
Status: Completed | Type: Observational
Sponsor: Rottapharm Spain (Industry)
Responsible Party: Sponsor
Other Study IDs: ESTROCALVI
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Menopause
Keywords: menopause; quality of life; soy isoflavones; magnolia extract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- isoflavones combined with magnolia: A food supplement containing soy isoflavones, lactobacillus sporogenous, Ca,vitamin D3, magnesium and magnolia extract will be administered once a day during 12 weeks.
  Interventions: Dietary Supplement: isoflavones combined with magnolia

INTERVENTIONS:
Dietary Supplement: isoflavones combined with magnolia — 1 tablet/day duration: 12 weeks
  Other Names: Estromineral Serena

SUMMARY:
In menopause, the vasomotor symptomatology, accompanied or less by affective and behavioural symptoms, globally worsens the quality of daily life.

The improvement of the quality could be reached with adequate food supplements, named phytoestrogens, in particular Soy Isoflavones (SI), which are natural substances with estrogen-like and estrogen-antagonistic activity, which are active in the control of menopausal vasomotor symptoms. Besides, combined with magnolia extract it could improve the psychological symptomatology also improving the quality of life.

DETAILED DESCRIPTION:
Multicenter, observational, prospective, longitudinal study of clinical practice conducted in 10 gynecological centers.

The study will be conducted in patients with typical mild to moderate vasomotor symptoms and psycho symptoms such as mood disorders, or sleep, anxiety / depression, which do not require specific drug treatment.

Quality of life will be analyzed by the scale of Cervantes.

ELIGIBILITY:
Inclusion Criteria:

* Women with at least 12 months of amenorrhea
* Presence of 1 or more vasomotor symptoms as hot flushing, nocturnal sweating or palpitations
* One or more psychological symptoms as insomnia, irritability, anxiety, depressed mood. Also with concomitant symptoms of sexual area as reduction of libido and vaginal dryness.
* Women must give the informed consent

Exclusion Criteria:

* clinical history of medical or surgical pathologies that could affect the results of the study, including serious cardiovascular, metabolic, kidney or liver diseases
* Patients with the habit of eating soy foods or dietary supplements with soy extract
* patients diagnosed with breast or uterine mass (neoplasia hormone sensitive)
* patients that were treated with estrogens (HRT or phytoestrogens)in the 2 months before the beginning of the study.
* patients with treatment with antibiotics, antidepressant and/or anxiolytic products

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will be conducted in patients with typical mild to mderate vasomotor symptoms and psycho symptoms such as mood changes, or sleep, anxiety / depression, which do not require specific drug treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
the quality of life measured by the scale of Cervantes | baseline and 12 weeks
  The Cervantes scale is a Spanish validated questionnaire specific for measure the quality of life in menopausal women

SECONDARY OUTCOMES:
Clinical changes in vasomotor symptomatology | baseline, 2, 4, 8 and 12 weeks
  In a semiquantitative scale of intensity the vasomotor, psychological and sexual symptomatology will be evaluated in each visit

CONTACTS AND LOCATIONS:
Overall Officials: Anna Anguera, MD, PhD, Study Director — Rottapharm S.L.; Rafael Sánchez-Borrego, MD, Principal Investigator — Centro Médico Teknon
Locations (10):
- Spain (10):
  - Somdex S.L., Barcelona, Barcelona
  - Centro Médico Teknon, Barcelona, Barcelona
  - Surgery of Dr. Sánchez Muñoz, Ciudad Real, Ciudad Real
  - Gabinete Médico Velazquez, Madrid, Madrid
  - Clínica ginecológica Cecchini, Oviedo, Oviedo
  - Instituto Sevillano de Ginecología y Obstetricia, Seville, Sevilla
  - Surgery of Dr. Mahiques, Valencia, Valencia
  - Surgery of Dr. Raga, Valencia, Valencia
  - Grupo hospitalario Quirón, Erandio, Vizcaya
  - Centro Ginecológico Dr. García Pérez-Llantada SL, Zaragoza, Zaragoza